CLINICAL TRIAL: NCT00419172
Title: A Phase I, Single Center, Open-label, One-sequence Cross-over Study to Investigate the Effect of a Potent Inducer Rifampicin on the Pharmacokinetics of Deferasirox in Healthy Volunteers
Brief Title: Effect of a Potent Inducer Rifampicin on the Pharmacokinetics of Deferasirox in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CICL670A2127
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Deferasirox; Exjade; ICL670; Rifampicin; Healthy, Volunteers
MeSH Terms: interventions — Deferasirox; Rifampin

INTERVENTIONS:
Drug: Deferasirox
Drug: Rifampicin

SUMMARY:
The study will consist of two open-label periods, a Treatment Period I (deferasirox) and a Treatment Period II (rifampicin+deferasirox). At least 18 subjects are expected to complete both treatment periods as per protocol. For all subjects, in addition to the two treatment periods, there will be a 21 day screening period, one baseline evaluation (the day preceding deferasirox administration in Treatment Period I), and an end-of-study evaluation (EOS). Study subjects will be required to remain in the unit from Day -1 until Day 17. EOS evaluation (final safety assessment) will be performed 7-10 days after the last dose of rifampicin.

ELIGIBILITY:
Inclusion criteria

1. Able and willing to provide written informed consent prior to study participation
2. Male subjects from 18 - 45 years of age in good health and no evidence of iron deficiency. Subjects of reproductive potential must use barrier contraception throughout the trial.
3. Able to communicate well with the investigator and comply with the requirements of the study
4. Subjects must have a body mass index (BMI) between 18 and 33.
5. Serum ferritin value ≥20 ng/mL and transferrin saturation (Iron/TIBC) ≥15% at screening

Exclusion criteria

1. History or presence of impaired renal function
2. Abnormal serum electrolytes (e.g. sodium, potassium, chloride, or bicarbonate), magnesium and calcium
3. Evidence of urinary obstruction or difficulty in voiding at screening
4. Anemia (defined as hemoglobin < 13 g/dL)
5. A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result at screening
6. Subjects with a known history of HIV seropositivity or history of immunocompromise
7. A past medical history of any ECG abnormalities or a family history of a prolonged QT-interval syndrome
8. Donation or loss of 400 mL blood or more within 12 weeks prior to dosing
9. Smokers (use of tobacco products in the previous 3 months). * Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2007-01

PRIMARY OUTCOMES:
Evaluate the effect of rifampicin on pharmacokinetics after single dose administration of deferasirox

SECONDARY OUTCOMES:
Assess the safety and tolerability of concomitant administration of rifampicin and deferasirox

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis